CLINICAL TRIAL: NCT04289610
Title: Evaluation of the Effectiveness of Transcutaneous Pulse Radiofrequency Treatment in Subacromial Impingement Syndrome Patients
Brief Title: Transcutaneous Pulse Radiofrequency Treatment for Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ayça Utkan Karasu, medical doctor, principal investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Gazi University PMR
Record Dates: First submitted 2020-02-12; First posted 2020-02-28 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Shoulder Pain; Transcutaneous radiofrequency treatment; Ultrasound
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Sham Comparator): In this group a pair of TCPRF electrodes will be applied to the painful shoulder at six standardized sites for 2 minutes each (approximately a total of 15 minutes). The device is not going to be activated in the control group. The device will be set at 0 V. TCPRF treatment is going to be applied for one session.
  Interventions: Device: Transcutaneous pulse radiofrequency therapy
- Study Group (Active Comparator): A pair of TCPRF electrodes will be applied to the painful shoulder at six standardized sites for 2 minutes each (approximately a total of 15 minutes). It will be activated in the study group. In the study group device will be set at 80 V, every pulse will continue for 10 milliseconds and 5 pulses per second. TCPRF treatment is going to be applied for one session in both groups.
  Interventions: Device: Transcutaneous pulse radiofrequency therapy

INTERVENTIONS:
Device: Transcutaneous pulse radiofrequency therapy — Transcutaneous pulse radiofrequency therapy (TCPRF) is a painless and outpatient physiotherapy modality

SUMMARY:
Shoulder pain is the most common musculoskeletal problem after low back and neck pain. Subacromial impingement syndrome is one of the most common diseases that causes shoulder pain. Many methods are used to reduce pain and accelerate functional rehabilitation in patients with shoulder pain. Transcutaneous pulse radiofrequency therapy (TCPRF) is a needle-free, painless, and outpatient physical therapy modality that can be used to treat shoulder impingement syndrome. Acromio-humeral distance and supraspinatus tendon thickness measurements with ultrasound are reliable and effective methods to diagnose subacromial impingement syndrome. Although there are previous studies investigating the effectiveness of TCPRF treatment in patients with shoulder pain, there are no studies evaluating the effectiveness of treatment with ultrasound examination. In this study, the investigators aimed to show the effect of TCPRF treatment on pain, range of motion, functional status and ultrasound findings in subacromial impingement syndrome.

DETAILED DESCRIPTION:
Shoulder pain is the most common musculoskeletal problem after low back and neck pain. It has negative socioeconomic effects on patient's daily life (1). Subacromial impingement syndrome is one of the most common diseases of the shoulder and seen in 44-65% of patients who consult a doctor with shoulder pain. This syndrome spectrum includes supraspinatus tendon partial tears, supraspinatus tendinitis, calcific tendinitis and subacromial bursitis. Many treatments are used to reduce pain and accelerate functional rehabilitation in patients with shoulder pain. These treatments include analgesic physical therapy agents (superficial hot and cold applications, deep heaters, diadynamic currents, transcutaneous electrical stimulation, interferential current, short wave diathermy), therapeutic exercises, massage, functional electrical stimulation, acupuncture, analgesics, non-steroid anti-inflammatory drugs, oral steroids and steroid injections. Transcutaneous pulse radiofrequency therapy (TCPRF) is a painless and outpatient physiotherapy modality that does not require any anesthesia or sedation. TCRPF can also be used in some other painful conditions of the chin, neck, lower back, wrist, knee, elbow and ankle regions. Ultrasound measurement of acromio-humeral distance and supraspinatus tendon thickness are reliable and effective methods for demonstrating subacromial impingement syndrome. Although there have been previous studies investigating the effectiveness of TCPRF treatment in patients with shoulder pain, the number of these studies are insufficient. In addition, there are no studies evaluating the effectiveness of treatment by ultrasound examination. In this study, the investigators aimed to evaluate the effect of TCPRF treatment on pain, range of motion and functional status in subacromial impingement syndrome patients by means of clinical and ultrasound findings.

The study will be conducted between January 2020 and January 2021 at Gazi University Faculty of Medicine, Department of Physical Medicine and Rehabilitation. Fifty patients with subacromial impingement syndrome are planned to be recruited for the study.

The patients included in the study will be randomized into two groups with a computer program. In order to comply with the double-blind study protocol, the researcher performing the randomization of the patients will not participate in the treatment and evaluation processes. Demographic data of patients will be recorded at the beginning of the study. Therapeutic exercises and nonsteroidal anti-inflammatory drug therapy will be initiated to all patients. Detailed shoulder joint range of motion examination, visual analog scale, shoulder pain and disability index, quality of life scale (SF-36), shoulder ultrasound examination for acromio-humeral distance and supraspinatus tendon thickness measurements will be performed before and after treatment (Basal, 1st, 4th and 12th weeks). A pair of TCPRF electrodes will be applied to the painful shoulder at six standardized sites for 2 minutes each (approximately a total of 15 minutes). The device is not going to be activated in the control group. It will be activated in the study group. In the study group device will be set at 80 V, every pulse will continue for 10 milliseconds and 5 pulses per second. In the control group the device will be set at 0 V. TCPRF treatment is going to be applied for one session in both groups. During the three-month follow-up period, therapeutic exercises and as long as it is considered necessary nonsteroidal anti-inflammatory drugs will be continued in both groups.

ELIGIBILITY:
Inclusion Criteria:

* 18- 65 years of age
* Having (chronic) shoulder pain for more than 3 months
* No treatment for shoulder pain (physical therapy, joint area injection, radiofrequency treatment) in the past 3 months

Exclusion Criteria:

* Systemic rheumatic diseases

  * Malignancy, acute infections Adhesive capsulitis
  * Bicipital tendinitis
  * Supraspinatus tendon full-thickness rupture
  * Those who have undergone surgery for shoulders and neck
  * Pace maker
  * Pregnant women Those with cervical radiculopathy
  * Those who do not agree to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
The effect of transcutaneous pulsed radiofrequency (TCPRF) treatment on shoulder pain in subacromial impingement syndrome. | Change from baseline VAS at 1st week, 4th week and 12th week.
  Shoulder pain will be assessed by visual analog scale (VAS). A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain. Two extreme definitions of pain (0: no pain, 10: The most powerfull pain one can exprience) are written on both ends of a 100 mm line and the patient is asked to indicate where his condition is appropriate by drawing a line or by marking or pointing on this line.
The effect of transcutaneous pulsed radiofrequency (TCPRF) treatment on shoulder range of motion in subacromial impingement syndrome. | Change from baseline shoulder range of motion at 1st week, 4th week and 12th week.
  Shoulder range of motion will be assessed by goniometer. A goniometer is an instrument that measures range of motion joint angles (degree) of the body . A goniometer will be used to evaluate shoulder joints.
The effect of transcutaneous pulsed radiofrequency (TCPRF) treatment on shoulder disability in subacromial impingement syndrome. | Change from baseline shoulder disability at 1st week, 4th week and 12th week.
  Shoulder disability will be assessed by shoulder pain and disability index (SPADI). SPADI is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The patient is asked to score how much difficulty he had during physical activities in the past week (zero means no difficulty, ten means unable to do the activity without help). Total score changes between 0 to 130. Zero defines no difficulty and 130 defines maximum disability.

SECONDARY OUTCOMES:
Measurement of Acromiohumoral Distance | Change from baseline acromiohumoral distance at 1st week, 4th week and 12th week.
  Acromiohumoral distance will be evaluated with ultrasound. Measurements will be defined as milimeters.
Assessment of Quality of life (QOL) | Change from baseline Assessment of Quality of life (QOL) at 1st week, 4th week and 12th week.
  Short form 36 Health Survey Questionnaire (SF-36) ill be used for QOL assessment. The SF-36 is a 36-item self-report measure of health-related quality of life and it is a reliable and valid questionnaire for musculoskeletal diseases. It has eight subscales measuring different domains of health-related quality of life: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. Two component scores are derived from the eight subscales: a physical and a mental health component score. The SF-36 also includes a single item that assesses perceived change in health status over the past year. The lower the score the more disability. Higher scores on all subscales represent better health and functioning.
Measurement of Supraspinatus Tendon Thickness | Change from baseline supraspinatus tendon thickness at 1st week, 4th week and 12th week.
  Supraspinatus tendon thickness will be evaluated with ultrasound. Measurements will be defined as milimeters.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Medical School, Physical Medicine and Rehabilitation Department, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
there is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Result] Taverner M, Loughnan T. Transcutaneous pulsed radiofrequency treatment for patients with shoulder pain booked for surgery: a double-blind, randomized controlled trial. Pain Pract. 2014 Feb;14(2):101-8. doi: 10.1111/papr.12059. Epub 2013 Apr 8. PMID 23560519
- [Result] Kul A, Ugur M. Comparison of the Efficacy of Conventional Physical Therapy Modalities and Kinesio Taping Treatments in Shoulder Impingement Syndrome. Eurasian J Med. 2019 Jun;51(2):139-144. doi: 10.5152/eurasianjmed.2018.17421. Epub 2018 Nov 30. PMID 31258353
- [Result] Taverner MG, Ward TL, Loughnan TE. Transcutaneous pulsed radiofrequency treatment in patients with painful knee awaiting total knee joint replacement. Clin J Pain. 2010 Jun;26(5):429-32. doi: 10.1097/AJP.0b013e3181d92a87. PMID 20473051
- [Result] McCreesh KM, Anjum S, Crotty JM, Lewis JS. Ultrasound measures of supraspinatus tendon thickness and acromiohumeral distance in rotator cuff tendinopathy are reliable. J Clin Ultrasound. 2016 Mar-Apr;44(3):159-66. doi: 10.1002/jcu.22318. Epub 2015 Dec 15. PMID 26666736